CLINICAL TRIAL: NCT01919099
Title: Natural History Study of the Complications Associated With Allogeneic Hematopoietic Stem Cell Transplantations
Brief Title: Study of the Complications Associated With Certain Stem Cell Transplants
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130177; 13-I-0177
Record Dates: First submitted 2013-08-07; First posted 2013-08-08 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Post-Transplant Infections; Post-Transplant Renal Insufficiency; Post-Transplant Pulmonary Complications
Keywords: Post-Transplant Infection; Post-Transplant Bacteremia; Post-Transplant Virus; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-transplant: Patients receiving allogenic stem cell transplants at the NIH CC

SUMMARY:
Background:

- The National Institutes of Health (NIH) performs up to 100 allogenic stem cell transplants (allo-HSCT) each year. Many studies already look at different problems that can follow a transplant. But there are many types of transplants, diseases, responses, and treatments. An organized study of this information could help researchers learn more about how often transplant complications occur and what problems they cause. It could also lead to ideas for future research. This study will focus on complications thought to be the most significant.

Objectives:

- To gather information on the complications that may occur after an allo-HSCT.

Eligibility:

- People over 2 years of age currently enrolled in an allo-HSCT study at NIH.

Design:

* Visits for this study will be scheduled along with primary study visits. The number of visits will depend on the primary study schedule.
* At each visit, participants will answer questions and take physical exams.
* The same questions and physical exams will continue for as long as they are in the primary study.
* In between visits, researchers might call participants to discuss their health. They may also discuss the cases with the primary study doctors and other doctors. Primary transplant study doctors will make treatment decisions.
* When participation in the primary transplant study ends, participation in this study will also end.

DETAILED DESCRIPTION:
Between 80 and 100 allogeneic stem cell transplants (allo-HSCT) are performed every year at the NIH to treat a variety of malignant and nonmalignant conditions. The current transplant protocols at the NIH focus on research regarding the response of the underlying disease, the development of graft versus host disease (GVHD) as well as the feasibility and safety of a variety of transplant strategies. Many clinically significant complications are considered to be part of the transplant process and are not studied systematically. Even when they are studied, the diverse institute-based protocols differ on the range of complications captured and the amount of information collected on them. This leads to knowledge gaps regarding the incidence and risk factors for complications in the various protocols.

This exploratory natural history study involves a prospective review of the medical records of patients actively enrolled in allo-HSCT protocols at the NIH. The study will focus on infections and a subset of noninfectious complications identified by the transplant community as significant causes of morbidity, mortality and cost. The cost data captured in this study will be the cost consumed by the Clinical Center. This study does not require any sample collection and will consist merely of data collection and optional periodic patient examinations that will be performed in conjunction with those already scheduled by the original transplant protocol. The prospective collection of clinical data and information available in the medical record will allow us to determine the rates of a number of complications in different protocols. At the completion of the study, it is expected the investigators will be able to generate preliminary hypotheses regarding risk factors for infection and noninfectious complications, the impact of complications on transplant costs and the correlation between laboratory immune reconstitution (usually determined by each transplant protocol in a variety of ways and functional immune reconstitution (frequency of infections).

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects over the age of 2 that are actively enrolled in an allo-HSCT protocol at any NIH institute will be eligible to participate in this study regardless of gender or medical condition. Patients may be consented prior to and up to a week after receiving the stem cells (Day 0 of transplant).

EXCLUSION CRITERIA:

Subjects with any condition that, in the opinion of the investigator, contraindicates participation in the study will be excluded.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From NIH transplant protocols
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-07-31 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2017-08-24 (Actual)

PRIMARY OUTCOMES:
Characterize the infectious and noninfectious complications associated with allo-HSCT, including incidence, clinical course, cost to the Clinical Center and distribution within each NIH intramural transplant protocol | Every few years or as requested by the clinical center or investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Christa S Zerbe, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] De Pauw B, Walsh TJ, Donnelly JP, Stevens DA, Edwards JE, Calandra T, Pappas PG, Maertens J, Lortholary O, Kauffman CA, Denning DW, Patterson TF, Maschmeyer G, Bille J, Dismukes WE, Herbrecht R, Hope WW, Kibbler CC, Kullberg BJ, Marr KA, Munoz P, Odds FC, Perfect JR, Restrepo A, Ruhnke M, Segal BH, Sobel JD, Sorrell TC, Viscoli C, Wingard JR, Zaoutis T, Bennett JE; European Organization for Research and Treatment of Cancer/Invasive Fungal Infections Cooperative Group; National Institute of Allergy and Infectious Diseases Mycoses Study Group (EORTC/MSG) Consensus Group. Revised definitions of invasive fungal disease from the European Organization for Research and Treatment of Cancer/Invasive Fungal Infections Cooperative Group and the National Institute of Allergy and Infectious Diseases Mycoses Study Group (EORTC/MSG) Consensus Group. Clin Infect Dis. 2008 Jun 15;46(12):1813-21. doi: 10.1086/588660. PMID 18462102
- [Background] Seo S, Campbell AP, Xie H, Chien JW, Leisenring WM, Englund JA, Boeckh M. Outcome of respiratory syncytial virus lower respiratory tract disease in hematopoietic cell transplant recipients receiving aerosolized ribavirin: significance of stem cell source and oxygen requirement. Biol Blood Marrow Transplant. 2013 Apr;19(4):589-96. doi: 10.1016/j.bbmt.2012.12.019. Epub 2013 Jan 5. PMID 23298855
- [Background] Azoulay E, Bergeron A, Chevret S, Bele N, Schlemmer B, Menotti J. Polymerase chain reaction for diagnosing pneumocystis pneumonia in non-HIV immunocompromised patients with pulmonary infiltrates. Chest. 2009 Mar;135(3):655-661. doi: 10.1378/chest.08-1309. PMID 19265086
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-I-0177.html